CLINICAL TRIAL: NCT05047458
Title: A Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACH-0145228 in Healthy Volunteers
Brief Title: A Study of Single-dose ALXN2050 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ACH228-001; ACTRN12617001521314 (Other: Australian New Zealand Clinical Trials Registry); U1111-1203-1371 (Other: Universal Trial Number)
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Factor D Inhibitor; Complement; ALXN2050; ACH-0145228; Pharmacokinetics; Pharmacodynamics; Safety
MeSH Terms: interventions — rhoA GTP-Binding Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1: 40 mg ALXN2050/Placebo (Experimental): Participants randomized to receive ALXN2050 or placebo on Day 1.
  Interventions: Drug: ALXN2050; Drug: Placebo
- Cohort 2: 80 mg ALXN2050/Placebo (Experimental): Participants randomized to receive ALXN2050 or placebo on Day 1.
  Interventions: Drug: ALXN2050; Drug: Placebo
- Cohort 3: 120 mg ALXN2050/Placebo (Experimental): Participants randomized to receive ALXN2050 or placebo on Day 1.
  Interventions: Drug: ALXN2050; Drug: Placebo

INTERVENTIONS:
Drug: ALXN2050 — Powder-in-capsule (PIC).
  Other Names: ACH-0145228 (formerly); ACH-5228
Drug: Placebo — PIC.

SUMMARY:
This was a phase 1, first-in-human, single-center, randomized, double-blind (participants and investigator blind, sponsor open) placebo-controlled, single-ascending dose study of ACH-0145228 (ALXN2050) conducted in healthy adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy was defined as having no clinically relevant abnormalities identified by a detailed medical history, physical examination, blood pressure and heart rate measurements, 12-lead ECG, and clinical laboratory tests.
* Had a body mass index of 18 to 30 kilograms (kg)/meter squared with a minimum body weight of 50 kg.
* Female participant of nonchildbearing potential.
* Male participant agreed to abstinence or use of a highly effective form of contraception.

Key Exclusion Criteria:

* Had a history or clinically relevant evidence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* Had any condition possibly affecting drug absorption.
* Had a body temperature greater than or equal to 38°Celsius on Day -1 or Day 1, Hour 0; had a history of febrile illness, or other evidence of infection, within 14 days prior to first study drug administration.
* Had a positive urine drug screen at Screening or Day -1; was a current tobacco/nicotine user or smoker; had consumed any alcohol within 72 hours before first study drug administration or had a history of regular alcohol consumption within 6 months of Screening.
* Had participated in a clinical study within 30 days prior to first study drug administration
* Had clinically significant laboratory abnormalities,
* Had donated blood or lost more than 500 milliliters of blood within 3 months prior to first study drug administration; had received a blood transfusion or blood products within 6 months prior to first study drug administration.
* Had a clinically significant history of drug allergy.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Number Of Participants Experiencing Serious Adverse Events | Day 1 through Day 42
Number Of Participants Experiencing Grade 3 Or 4 Adverse Events (AEs) | Day 1 through Day 42
Number Of Participants Experiencing AEs Leading To Discontinuation From The Study | Day 1 through Day 42
Number Of Participants Experiencing Grade 3 Or 4 Laboratory Abnormalities | Day 1 through Day 42
Number Of Participants Experiencing Treatment-emergent Vital Signs, Physical Examination Results, And Electrocardiogram (ECG) Abnormalities | Day 1 through Day 42

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) Of ALXN2050 | Up to 144 hours postdose
Time To Reach The Maximum Plasma Concentration (Tmax) Of ALXN2050 | Up to 144 hours postdose
Area Under The Plasma Concentration-time Curve Extrapolated To Infinity (AUC0-inf) Of ALXN2050 | Up to 144 hours postdose
Alternative Pathway (AP) Activity As Measured By Wieslab Assay | Up to 144 hours postdose
Plasma Bb Fragment Of Complement Factor B Concentration Over Time | Up to 144 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes